CLINICAL TRIAL: NCT03546296
Title: Dietary Factors and Risk of Gallbladder Carcinoma in China
Acronym: DRGBC001
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yingbin Liu, MD, PhD, FACS (Other)
Collaborators: The First Hospital of Jilin University (Other); Shanghai Zhongshan Hosiptal (Unknown); The First Affiliated Hospital of Bengbu Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Jining Medical University (Other); The Affiliated Hospital of Tianjin Medical University (Unknown); The first affiliated hospital of Zhongshan university (Unknown)
Responsible Party: Sponsor-Investigator, Yingbin Liu, MD, PhD, FACS, vice-president，Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: GBC2017
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Dietary Habits
Keywords: Dietary Exposure; gallbladder carcinoma
MeSH Terms: conditions — Feeding Behavior; Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will obtain the blood and urine samples for further analysis of metabolomics studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to see how people's diets, other aspects of their lifestyles affect their chances of getting gallbladder carcinoma in China. This survey will enroll 100 patients who have had gallbladder carcinoma，as well as controls with gallstones. The investigators will compare these two groups of subjects to see what factors may lead to gallbladder carcinoma.

DETAILED DESCRIPTION:
The investigators will conduct a case-control study in 10 hospitals from China. Cases will be the patients with newly-diagnosed gallbladder carcinoma. The controls will be matched （1：1）by sex，race and age which will be selected from the patients receiving cholecystectomy due to gallstones from the same hospital with the cases.

There will be 100 cases with gallbladder carcinoma, 100 controls. The investigators will interview participants about known and potential risk factors for gallbladder carcinoma and obtain information on diet. The investigators will obtain the blood and urine samples for further analysis of metabolomics studies. The investigators will use logistic regression to determine odds ratios for disease with various exposures.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with gallbladder carcinoma by imaging tests (cases) Diagnosed with chronic cholecystitis by imaging tests (hospital controls)

Exclusion Criteria:

The pathology diagnosis and imaging does not matched Patients with other malignant tumors Patients with other severe systemic diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will conduct a case-control study in 11 hospitals from China. Cases will be the patients with newly-diagnosed gallbladder carcinoma. The hospital controls will be matched （1：1）by sex，race and age which will be selected from the patients receiving cholecystectomy due to gallstones from the same hospital with the cases. The community controls will be matched（1：1） by sex，race and age which will be selected from the same community with the cases.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the The demographic, reproductive, and lifestyle characteristics | 2017-2019
  Cases and controls were interviewed by one of three research assistants with a standard questionnaire to elicit information about demographic, reproductive, and lifestyle characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China